CLINICAL TRIAL: NCT06325878
Title: Dissecting the Genetic Architecture of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: Genetic Architecture of Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: GEARCIDP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NEU2-OSS-2022-001
Record Dates: First submitted 2024-03-16; First posted 2024-03-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Keywords: Chronic Inflammatory Polyradiculoneuropathy; Polyneuropathy, Inflammatory Demyelinating, Chronic; Chronic Inflammatory Demyelinating Polyradiculoneuropathy; cidp
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Genome-Wide Association Study

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chronic inflammatory demyelinating polyneuropathy (CIDP) (Experimental): Single nucleotide polymorphisms (SNPs) of 1000 patients with chronic inflammatory demyelinating polyneuropathy will be genotyped using the Illumina Global Screening Array
  Interventions: Genetic: Genome-wide association study
- Control Subjects (Experimental): Single nucleotide polymorphisms (SNPs) of 2500 control subjects without chronic inflammatory demyelinating polyneuropathy will be genotyped using the Illumina Global Screening Array
  Interventions: Genetic: Genome-wide association study

INTERVENTIONS:
Genetic: Genome-wide association study — Alleles/haplotypes evidence through GWAS will be compared between patients with CIDP and control subjects without CIDP

SUMMARY:
The objective of this study is to characterize the genetic architecture of a large cohort of CIDP patients to evaluate whether specific alleles/haplotypes are implicated in the risk of CIDP, in its clinical and immunological variability, severity, therapeutic response, and association with diabetes and other autoimmune diseases. We will genotype >700,000 single nucleotide polymorphisms (SNPs) by using the Illumina Global Screening Array (GSA), of approximately 1000 patients with CIDP. About 3500 healthy controls from the Italian population have been already genotyped using GWAS from our genetic department. Alleles/haplotypes will be also compared between patients with typical CIDP and its variants, between CIDP patients with and without specific antibodies, between CIDP patients with and without comorbidities, between CIDP patients with low and high levels of disability and between CIDP patients with and without response to each individual treatment (IVIg, steroids, plasma exchange)

DETAILED DESCRIPTION:
1. Specific aim 1: Characterize the genetic architecture of CIDP by using a genome-wide association study (GWAS) approach in a large cohort of CIDP patients and healthy controls, thus defining the 1) Specific aim 1: Characterize the genetic architecture of CIDP by using a genome-wide association study (GWAS) approach in a large cohort of CIDP patients and healthy controls, thus defining the spectrum of single common variants or their combinations (in terms of haplotypes or risk score) predisposing to the disease.

   Hypothesis: The frequency of specific alleles/haplotypes in patients with CIDP is significantly different compared to that of the general population.

   Approach: We will genotype >700,000 single nucleotide polymorphisms (SNPs) by using the Illumina Global Screening Array (GSA), of approximately 1000 patients with CIDP. About 3500 healthy controls from the Italian population have been already genotyped using GWAS from our genetic department (Prof. Asselta, Humanitas Research Institute, Milan).
2. Specific aim 2: Explore the role of specific alleles/haplotypes in determining the clinical and immunological variability, severity, and therapeutic response of CIDP.

   Hypothesis: The genetic architecture of patients with typical CIDP is -at least in part- distinct from that of the CIDP variants; specific alleles/haplotypes associate with intermediate phenotypes, such as the presence of antibodies anti-NF155, anti-NF186, CNTN1, anti-gangliosides; Specific alleles/haplotypes correlate with severity and treatment-response of CIDP.

   Approach: Alleles/haplotypes evidence through GWAS will be compared between patients with typical CIDP and its variants, between CIDP patients with and without specific antibodies, between CIDP patients with low and high levels of disability and between CIDP patients with and without response to each individual treatment (IVIg, steroids, plasma exchange) in order to determine whether genetics play a role in determining these phenotypes.
3. Specific aim 3: Verify possible overlaps between CIDP and other autoimmune diseases.

Hypothesis: Alleles/haplotypes identified through GWAS play a role in the increased risk of diabetes and other autoimmune disease in CIDP.

Approach: Alleles/haplotypes evidence through GWAS will be compared between CIDP patients with and without diabetes mellitus, and with and without any other autoimmune diseases.

This is a multicenter, international, observational study where a large number of CIDP patients will be screened using GWAS. About 3500 healthy controls from the Italian population have been already genotyped using GWAS. Patients with a diagnosis of CIDP according to the current diagnostic criteria will be included. Patients with autoimmune nodopathies will be also included. Patients must give informed consent to participate. For all the patients, the diagnosis at enrollment will be revised by the coordinating Center, according to the European Academy of Neurology/Peripheral Nerve Society (EAN/PNS) diagnostic criteria.

All included patients will undergo a detailed clinical history including time of clinical onset, presence - distribution and date of onset of motor and sensory symptoms, ataxia, pain, tremor, cramps, fatigue, autonomic dysfunction, and cranial nerve involvement using a specific questionnaire. This information will be integrated with the data reported in the medical records. Disease course will be defined as progressive, relapsing or monophasic by the treating neurologist. The clinical evaluation at enrolment will include assessment of muscle strength using the Medical Research Council (MRC) sumscore on 12 muscles (range 0-60). Neurological disability will be evaluated at enrollment with the Inflammatory-Rash Overall Built Disability Scale (I-RODS), and the Inflammatory Neuropathy Cause and Treatment (INCAT) disability scale, while Quality of life (QoL) will be assessed with the EuroQol-5D-3L scale. Response to treatment will be defined as a subjective improvement that was objectively confirmed by I-RODS: + ≥ 4 centile points, or INCAT disability scale (≥ 1 point), or MRC sum score (0-60) (≥ 2-4 points), or grip strength using Martin Vigorimeter (≥ 8 -14 kPa).6 Results of previously performed examinations including cerebrospinal fluid (CSF) analysis, nerve ultrasound or brachial/lumbosacral plexus MR (magnetic resonance) examination and sural nerve biopsy, will be included when available. The results of nerve conduction studies performed during the course of the disease will be included. Sensory nerve conduction studies will be performed bilaterally in median, ulnar and sural nerves and included evaluation of sensory nerve action potential amplitude, distal latency and sensory conduction velocity. Motor nerve conduction studies will be also performed bilaterally in median, ulnar, common peroneal and tibial nerves and included distal and proximal compound muscle action potential amplitude and duration, motor conduction velocity, distal and proximal motor latency and in most patients F-wave latency. Abnormalities of motor and sensory nerve conduction studies consistent with demyelination will be defined according to the EAN/PNS criteria. In all the patients, the diagnosis at entry will be revised by the coordinating Center according to the above-mentioned diagnostic criteria.

Patient's data will be shared under pseudonymised form using the patients' code among the centres.

Enrollment in the study will be offered to all patients included in the Italian CIDP database. Enrollment will then be extended to other Italian and European centers

ELIGIBILITY:
Inclusion Criteria:

- Subject with a documented diagnosis of according to the EAN/PNS criteria

Exclusion Criteria:

* Subject with an alternative diagnosis for the neuropathy
* Subject without available nerve conduction studies or documented diagnosis of CIDP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
single nucleotide polymorphisms (SNPs) | 3 years
  Differences in single nucleotide polymorphisms (SNPs) between CIDP patients and controls

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Emiliano Doneddu, MD, Principal Investigator — Humanitas Research Institute
Locations (1):
- IRCCS Istituto Clinico Humanitas, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No